CLINICAL TRIAL: NCT03094468
Title: A Multicenter, Randomized, Double-blind, Parallel, Vehicle-controlled Study to Evaluate the Efficacy and Safety of P-3058 10% Nail Solution in the Treatment of Onychomycosis
Brief Title: Study to Evaluate the Efficacy and Safety of P-3058 Nail Solution in the Treatment of Onychomycosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Project development priorities changed
Sponsor: Polichem S.A. (Industry)
Collaborators: Almirall, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PM1328
Record Dates: First submitted 2017-03-21; First posted 2017-03-29 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Onychomycosis of Toenail
Keywords: terbinafine nail solution; nail fungal infection; topical antifungal drug

STUDY DESIGN:
Intervention Model Description: Vehicle-controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- P-3058 (Experimental)
  Interventions: Drug: P-3058 (terbinafine hydrochloride 10%)
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle of P-3058

INTERVENTIONS:
Drug: P-3058 (terbinafine hydrochloride 10%) — Patients will apply the P-3058 nail solution once weekly in a double blind fashion. The overall treatment phase is of 48 weeks.
  Arms: P-3058
Drug: Vehicle of P-3058 — Patients will apply the Vehicle of P-3058 once weekly in a double blind fashion. The overall treatment phase is of 48 weeks.
  Arms: Vehicle

SUMMARY:
The aim of this phase III study is to establish the efficacy and safety of P-3058 (terbinafine 10% nail solution) topically administered once weekly in patients with onychomycosis in comparison to the Vehicle in a double-blind fashion. The overall treatment period will be of 48 weeks.

DETAILED DESCRIPTION:
The study will consist of a screening phase, a treatment phase of 48 weeks and a 12-week follow-up. Patients affected by mild to-moderate distal lateral subungual onychomycosis (DLSO) on a target great toenail will be included in the study. Clinical as well as mycology assessments will be performed throughout the whole study. Safety will be monitored by recording any adverse event and evaluating local tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before starting any study related procedures.
* Patients aged 12 and older of any race.
* Males or females.
* Outpatients.
* Clinically diagnosed mild-to-moderate distal lateral subungual onychomycosis (DLSO) of at least one great toenail (the "target nail") at the Screening visit (V1).
* Patients with onychomycosis involving ≥ 20% to ≤ 50% of the area of the target great toenail.
* Patients with a positive KOH examination.
* Patients with positive culture for dermatophyte(s).
* Evidence of target great toenail growth reported by the patient defined as at least monthly nail clipping.

Exclusion Criteria:

* Woman who is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Patients with history of allergic reactions to terbinafine or its excipients.
* Use of any investigational drug/device or participation in a previous clinical trial within four weeks prior to Screening visit (V1).
* Patients using nail polish or other nail cosmetic product on the concerned nails from at least 24 hours prior to Screening visit (V1) until the end of the study.
* Use of systemic antifungal drugs in the 24 weeks prior to Screening visit (V1) or non-responsive to systemic antifungal therapy for onychomycosis.
* Nail application of topical antifungal drugs or device in the 4 weeks prior to Screening visit (V1).
* Presence of any nail infections other than dermatophyte.
* Presence of onychodystrophy that could interfere with clinical assessments.
* Presence of "yellow spikes" on the target nail.
* Presence of dermatophytoma on the target nail.
* Presence of nail thickness exceeding 2 mm.
* Patients with proximal subungual involvement (marker of immunosuppressed patient).
* Patients with severe plantar or moccasin tinea pedis (defined by blistering, pustules or inability to ambulate).
* Patients with nail abnormalities due to conditions like psoriasis, lichen planus, immune dysfunction, collagen-vascular diseases, peripheral vascular disease.
* Patients with life expectancy less than 2 years.
* Chemotherapy, immunosuppressive therapy in the 12 weeks prior to Screening visit (V1).
* Systemic corticosteroids, antimetabolites and immune-stimulants therapy in the 4 weeks prior to Screening visit (V1).
* HIV infection or any other immunodeficiency.
* Alcohol or substance abuse.
* Patients/parents (or legal guardian) unable to understand the procedures and purposes of the study.
* Any other condition that, in the opinion of the Investigator, would prevent the subject from effectively participating in the study, place the subject at risk or effect the assessment of efficacy and safety of the study medication.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Rate of complete cure at Week 60 | Baseline - Week 60
  Defined as composite of negative KOH microscopy and negative culture for dermatophytes and no residual clinical involvement (nail totally clear) of the target nail.

SECONDARY OUTCOMES:
Responder rate at Week 60 | Baseline - Week 60
  Defined as negative Potassium Hydroxide (KOH) microscopy and negative culture for dermatophytes and ≤ 10% residual involvement of the target toenail)
Mycological cure rate at Week 60 | Baseline - Week 60
  Defined as negative Potassium Hydroxide (KOH) microscopy and negative culture for dermatophytes of the target nail.

OTHER OUTCOMES:
Negative culture rate for dermatophytes of the target nail at Week 60 | Baseline - Week 60
Onychomycosis quality of life | Baseline - Week 48, Week 60
  The questionnaire ONYCHO (Toenail from Mapi Research Trust) will be administered at Week 0, at Week 48 and at Week 60 or at the discontinuation visit.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Caserini, MD, Study Director — Polichem SA
Locations (26):
- United States (21):
  - Polichem Investigation Site no 45, North Hollywood, California
  - Polichem Investigation Site no 5, Oceanside, California
  - Polichem Investigation Site no 39, San Diego, California
  - Polichem Investigation Site no 2, Hialeah, Florida
  - Polichem Investigation Site no 23, Jacksonville, Florida
  - Polichem Investigation Site no 22, Miami, Florida
  - Polichem Investigation Site no 52, Louisville, Kentucky
  - Polichem Investigation Site no 41, Portsmouth, New Hampshire
  - Polichem Investigation site no 1, New York, New York
  - Polichem Investigation Site no 44, Cincinnati, Ohio
  - Polichem Investigation Site no 40, Norman, Oklahoma
  - Polichem Investigation Site no 14, Oklahoma City, Oklahoma
  - Polichem Investigation Site no 10, Austin, Texas
  - Polichem Investigation Site no 11, Dallas, Texas
  - Polichem Investigation Site no 43, Dallas, Texas
  - Polichem Investigation Site no 6, Fort Worth, Texas
  - Polichem Investigation Site no 12, Houston, Texas
  - Polichem Investigation Site no 4, Houston, Texas
  - Polichem Investigation Site no 42, Pflugerville, Texas
  - Polichem Investigation Site no 53, San Antonio, Texas
  - Polichem Investigation Site no 54, San Antonio, Texas
- Canada (5):
  - Polichem Investigation site no 3, Calgary, Alberta
  - Polichem Investigation Site no 8, Edmonton, Alberta
  - Polichem Investigation Site no 13, Mississauga, Ontario
  - Polichem Investigation Site no 9, Richmond Hill, Ontario
  - Polichem Investigation Site no 7, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided